CLINICAL TRIAL: NCT02341729
Title: Evaluation of the Effects and Plasma Concentration of the Potent Platelet Inhibitor Ticagrelor, After Crushed and Non-crushed Intake, After Semi-urgent Coronary Bypass and in Patients After Cardiac Arrest.
Brief Title: Effects and Plasma Concentration of Ticagrelor, After Crushed and Non-crushed Intake, After Acute Coronary Syndrome
Acronym: ticagrelor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Intensievezorgen, Harlinde Peperstraete, Staff member ICU, University Hospital, Ghent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGO/2013/011
Record Dates: First submitted 2014-12-18; First posted 2015-01-19 (Estimated); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Acute Coronary Syndrome
Keywords: semi-urgent CABG; reanimation; ticagrelor; crushed tablet
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- starting with ticagrelor (Other): Patients, after CPR because of an ACS, will receive 2 crushed tablets of ticagrelor (180mg) through a gastric tube. After this dose twice a day 90mg is given for the duration of 1 year. The 1st blood sample is taken before administration. In total 10 blood samples are taken for determination of platelet aggregation and plasma concentrations.
  When patients receive a semi-urgent CABG, ticagrelor has been interrupted for 3 days. Postoperative the patients get crushed tablets of ticagrelor, the 1st dose will be 90mg, and every 12h 90mg is given, for the duration of 1 year. The 1st blood sample is taken before the 1st dose. In total 9 blood samples are taken for determination of platelet aggregation and plasma concentrations.
  Interventions: Drug: ticagrelor

INTERVENTIONS:
Drug: ticagrelor — crushed tablets and non-crushed tablets
  Other Names: Brilique

SUMMARY:
The first aim of the study is to prove that after starting the therapy with crushed tablets, the platelet inhibition will be as expected after starting therapy with intact tablets. Gurbel et al. showed that 100% of the patients on ticagrelor treatment have a decrease from baseline platelet aggregation of >10% 4 hours after last maintenance dose. So the investigators expect that after 3 days of treatment, all of our patients will have a closing time of more than 106seconds.

The investigators will observe two different clinical conditions of Acute Coronary Syndrome. First after semi-urgent coronary artery bypass graft (CABG) surgery, secondly in patients after cardiac arrest.

Both are clinical situations in which crushed tablets are needed to give. The second objective is to determine plasma concentrations of Ticagrelor and AR-C124910XX (active metabolite of ticagrelor) in these two patient populations after receiving 180mg or 90mg start-dose. Determination of plasma concentrations is done after protein precipitation, by using liquid chromatography with mass spectrometry detection. Measurements will be determined before intake (0h) and at 0,5; 1; 2; 4; 8; 24h and at day 4 +4h.7 The first 24h this will be a crushed tablet and 4 hours after the first intake at day 4 of therapy, this will be a non crushed tablet.

DETAILED DESCRIPTION:
This study is a single-centre, open-label, non-randomised longitudinal study in which the effect of ticagrelor, both crushed and non-crushed will be evaluated in two separate clinical conditions. The plasma concentrations after a crushed intake will be used to determine the maximum plasma concentration and time to achieve this maximum concentration.

50 patients of each condition:

Condition A: patients who received CPR because of cardiac arrest. A gastric tube is inserted. Subjects receive 2 crushed tablets of ticagrelor (180mg) with 10 ml water and a flush of 20 ml water. The first blood sample is taken before administration. The following samples are taken at 30minutes, 1, 2, 4, 8, 12, and 24h. The ninth sample is taken 24 hours after stopping sedation and 4h after administration of ticagrelor with 10 ml water and a flush of 20 ml water via nasogastric tube. The tenth sample is taken 4 days and 4hours after first intake of ticagrelor, this last sample is mostly after a non-crushed intake of ticagrelor (this depends on the neurological condition of the patient). Only the first dose is a loading dose of 180mg, hereafter a normal dose of 90mg is given.

At each blood sampling moment 1 or 2 samples are taken (see also flow chart). At time 0, 2, 4, 8, 12, 24h, 24h after sedation stop and at 4 days and 4hours after first intake of ticagrelor: a Platelet Function Analysis and an Aggreguide aggregometry is done. For each analysis 3,6ml of blood is needed, this makes a total of 28,8ml for the clotting analyses. At time 30min, 1, 2, 4, 8, 24h and 4 days and 4h; 4ml of blood is needed for the plasma concentration measurements, a total of 28ml.

Condition B: Patients in need of semi-urgent coronary bypass surgery, allowing interrupting the administration of ticagrelor 3 days before surgery. A nasogastric tube is inserted during surgery. On intensive care the patients will receive crushed tablets of ticagrelor with 10 ml water and a flush of 20 ml water via gastric tube, the first dose will be a loading dose. The first blood sample is taken just before surgery (weak effect of ticagrelor because administration has stopped 3 days). The following samples are taken at 30minutes, 1, 2, 4, 8, 12, and 24h. The ninth sample is taken 24 hours after stopping sedation and 4h after administration of ticagrelor with 10 ml water and a flush of 20 ml water via nasogastric tube. The tenth sample is taken 4 days and 4hours after first intake of ticagrelor, this last sample is mostly after a non-crushed intake of ticagrelor (this depends on the neurological condition of the patient). Only the first dose is a loading dose of 180mg, hereafter a normal dose of 90mg is given.

At each blood sampling moment 1 or 2 samples are taken (see also flow chart). At time 0, 2, 4, 8, 12, 24h, 24h after sedation stop and at 4 days and 4hours after first intake of ticagrelor: a Platelet Function Analysis and an Aggreguide aggregometry is done. For each analysis 3,6ml of blood is needed, this makes a total of 25,2ml for the clotting analyses. At time 30min, 1, 2, 4, 8, 24h and 4 days and 4h; 4ml of blood is needed for the plasma concentration measurements, a total of 28ml.

ELIGIBILITY:
Inclusion Criteria:

* Subject with an acute myocardial infarction with ST elevation
* Subject with an acute myocardial infarction without ST elevation
* Subject with unstable angina (progressive angina during past 2 weeks, negative cardiac markers, Trop T < 0,014μg/l
* First time of taking Brilique
* ≥ 18 years
* Possibility to take a blood sample before administration of Brilique
* Signed Informed Consent, signed by subject or authorized representative, able and willing to provide written informed consent for study participation

Exclusion Criteria:

* Active haemorrhage
* Moderate or severe liver failure with coagulopathy
* Pregnancy and lactation
* A history of an intra cerebral haemorrhage
* Patient is HIV positive and treated with Ritonavir and /or Atazanavir
* Patient treated with vitamin K antagonist or with a new oral anti coagulant
* Hypersensitivity to ticagrelor or any of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Platelet Function Analysis (closing time) and Aggreguide aggregometry (clotting analyses) | 5 days
  The first aim of the study is to prove that after starting the therapy with crushed tablets, the platelet inhibition will be as expected after starting therapy with intact tablets.
Plasma concentration measurements : plasma concentrations (using liquid chromatography with mass spectrometry detection) | 5 days
  The second objective is to determine plasma concentrations of Ticagrelor and AR-C124910XX in these two patient populations after receiving 180mg or 90mg start-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Harlinde Peperstraete, MD, Principal Investigator — Staff member at Ghent University Hospital
Locations (1):
- Intensive Care Unit, Ghent University Hospital, Ghent, Belgium

REFERENCES:
- [Derived] Duvillier L, Verhaege C, Devreese KMJ, Gevaert S, Peperstraete H. Evaluation of the effects and plasma concentration of the platelet inhibitor ticagrelor, after crushed and non-crushed intake, after cardiac arrest and after semi-urgent coronary artery bypass surgery. Acta Cardiol. 2024 Sep;79(7):805-812. doi: 10.1080/00015385.2024.2409521. Epub 2024 Oct 8. PMID 39377148